CLINICAL TRIAL: NCT03818997
Title: DKN-01/Atezolizumab as Second Line Treatment of biliarY Tract Cancer and in combiNAtion or Not With Paclitaxel as Second Line treatMent of esophagogastrIC Cancer: a Multi-center Phase II Trial
Brief Title: Combination of Targeted and Immunotherapy for Advanced Biliary Tract and Esophagogastric Gastric Cancer
Acronym: DYNAMIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry); Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1741-GITCG
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Cancer; Biliary Tract Cancer; GastroEsophageal Cancer; Hepatobiliary Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms; Biliary Tract Neoplasms | interventions — atezolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- BTC Cohort (Experimental): Patient in BTC cohort will receive immune therapy and DKN-01 IV until PD
  Interventions: Drug: DKN-01; Drug: Atezolizumab
- EGC cohort: DKN-01/atezolizumab + paclitaxel (Arm 1) (Experimental): Patient randomized in the EGC Arm 1 will receive immune therapy, DKN-01 and chemotherapy intravenously (IV) until PD.
  Interventions: Drug: DKN-01; Drug: Atezolizumab; Drug: Paclitaxel
- EGC cohort: DKN-01/atezolizumab without paclitaxel (Arm 2) (Experimental): Patient randomized in the EGC Arm 2 will receive immune therapy and DKN-01 IV until PD
  Interventions: Drug: DKN-01; Drug: Atezolizumab

INTERVENTIONS:
Drug: DKN-01 — Patient will receive DKN-01 300 mg IV every 2 weeks
Drug: Atezolizumab — Patient will receive Atezolizumab 840 mg IV every 2 weeks until PD
  Other Names: Tecentriq
Drug: Paclitaxel — Patient will receive Paclitaxel 80 mg/m2 IV on day 1, 8 and 15 of a 28 day cycle until PD
  Arms: EGC cohort: DKN-01/atezolizumab + paclitaxel (Arm 1)

SUMMARY:
In this study, non-operable esophagogastric adenocarcinoma cancer patients or non-operable biliary cancer patients whose cancer progressed/spread/got worse after first line treatment will be treated with or without immunotherapy and chemotherapy. This study will take place in several countries across Europe. One hundred twenty-three (123) patients will be invited to participate in this study

Biliary tract cancer (BTC), is a form of cancer that start in your bile ducts, a series of tubes that runs from the liver to the small intestines. It is not know yet the exact cause of BTC. For patients who have advanced or metastatic BTC (where surgery is not possible), chemotherapy is the first option for treatment. Chemotherapy with cisplatin and gemcitabine (CisGem) is the current standard of care.

Esophagogastric cancer (EGC) is cancer that occurs in the esophagus, a long hollow tube that runs from your throat to your stomach. The accumulating abnormal cells form a tumor in the esophagus that can grow to invade nearby structures and spread to other parts of the body. It's thought that chronic irritation of your esophagus may contribute to the changes that cause esophageal cancer.

The purpose of this study is to look at the risks and benefits of combining DKN-01 and atezolizumab (humanized monoclonal antibody) with or without paclitaxel (chemotherapy). Immune therapy boosts the body's natural defenses to fight cancer. It uses specific products made either by participants' body or in a laboratory to improve, target or restore immune system function and control or stop cancer. Atezolizumab is such an "immunotherapy" drug. DKN-01 is another new type of drug (humanized monoclonal antibody) in development as anticancer agent. Paclitaxel is a commonly-used chemotherapy drug of the class of taxanes used to treat a number of cancer types, it stimulates the cell to die or to stop the cell from dividing into two new cells.The idea behind combining these drugs is linked to targeting the immune system to attack the tumor. Combining immune and chemotherapy has already demonstrated clinical activity in relapsed (return of the disease)/refractory (not responding to treatment) esophagogastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of metastatic or locally unresectable adenocarcinoma of the biliary tract or esophagogastric adenocarcinoma.
* Measurable disease by CT/MRI (RECIST 1.1) within 28 days of randomization/enrollment
* Male and female subjects of age ≥18 years
* Performance status ECOG 0-1
* Life expectancy ≥ 4 months
* Normal 12-lead ECG (patients with abnormal ECG will be eligible if changes are not considered clinically significant by the local investigator)
* Adequate hematological function

  * Hemoglobin ≥ 9 g/dl (prior transfusions are allowed if they have been done ≥ 7 days before testing the Hb)
  * White blood cell (WBC) ≥ 3.0 x 109/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 75 x 109/L
* Adequate liver function: screening labs should be performed within 7 days prior to randomization/enrollment:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN), except subjects with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN.
  * ALT, AST & alkaline phosphatase ≤ 3 x ULN; ≤ 5 x ULN in case of liver/bone metastases
  * Serum albumin ≥ 2.5 g/dL
* Adequate renal function:

  o Estimated glomerular filtration rate (eGFR) according to MDRD should be > 50 ml/min
* Adequate coagulation:

  o International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants
* The following local treatment modalities are allowed within the rules described (provided there has been a full recovery):

  * Surgery: patients may have undergone a non-curative operation (i.e. R2 resection [with macroscopic residual disease] or palliative bypass surgery only), performed at least 28 days before randomization/enrollment. Patients who have previously undergone curative surgery, must have evidence of non-resectable and measurable disease relapse requiring systemic chemotherapy prior to study entry.
  * Radiotherapy: patients may have received prior radiotherapy (with or without radiosensitising low-dose chemotherapy) for localised disease. However, there must be clear evidence of disease progression post-treatment prior to inclusion in this study. The radiotherapy should have been finished at least 15 days prior to randomization/enrollment.
  * Photodynamic therapy (PDT) for localized disease only with no evidence of metastatic disease - patients may have received prior PDT, provided the patient has fully recovered and at least 28 days have elapsed since the PDT and there is clear evidence of disease progression at the local site or disease or at a new metastatic site.
  * Other previous localised treatments targeting intrahepatic lesions such as selective internal radiation therapy (SIRT), transarterial chemoembolisation (TACE) and radiofrequency ablation are allowed, provided the patient has finished it at leas 15 days prior to randomization/enrollment, with recovering.
* Asymptomatic subjects with known Central Nervous system (CNS) metastases are eligible, provided that all of the following criteria are met:

  * Measurable disease, per RECIST v1.1, must be present outside the CNS.
  * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
  * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
  * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to enrollment /randomization.
  * Any brain metastases must be stable for at least 6 months.
* Availability of 1 FFPE block (preferred) or if not available, minimum 15-20 freshly cut (≤ 7 days) unstained slides of tumor tissue (either from current or previous resection/biopsy) for biobanking/translational research if less tumor tissue available please contact the HQ study team.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures and agree to refrain from donating eggs, according the standard national guidelines during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomised partner
  * Sexual abstinence. Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Before patient enrollment, written informed consent must be given according to ICH/GCP, and national/local regulations.

Specific to BTC:

* Patients should have progressed after first line systemic therapy.
* If clinically indicated, adequate biliary drainage should have been performed, patient should have fully recovered.

Specific to advanced EGC:

•Patients who have progressed after first line therapy. HER2 positive patient should have received and progressed on trastuzumab therapy. In HER2 positive patient, neo/adjuvant therapy based on a platinum and a fluoropyrimidine could be considered a first line of therapy if the patient progressed within the first 3 months of completing it.

Note: patients who have undergone palliative treatment for obstruction or bleeding maybe eligible as long as they fulfill the above mentioned hematologic and biochemistry criteria.

* Weight must be stabilized in the last 4 weeks , as assessed by the investigator
* Taxanes, such as paclitaxel or docetaxel are only allowed in the curative setting (perioperative treatment) if received at least 12 months before enrollment/randomization.

Exclusion Criteria:

* Subjects with pleural effusion, pericardial effusion, or ascites with symptoms uncontrolled by medication or who requirere current drainage procedures (once monthly or more frequently).
* Leptomeningeal spread of disease.
* Patient is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks prior to enrollment
* Other concomitant or prior malignancy within the last 5 years, with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix.
* History of inflammatory bowel disease or any autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, type I diabetes mellitus, vasculitis, or glomerulonephritis
* Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
* Patients with controlled Type I diabetes mellitus on a stable insulin regimen are eligible.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  * Rash must cover less than 10% of body surface area.
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
  * Occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* History of radiation pneumonitis/fibrosis in the radiation field is permitted.
* Infections:

  * Signs or symptoms of infection or therapeutic use of antibiotics (except prophylactic antibiotics) within 2 weeks prior to randomization and severe infections within 4 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
  * Known or current evidence of HIV (test to be performed within 14 days of randomization)
  * Active or chronic hepatitis B or hepatitis C

    * Patients with past/resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. HBV DNA must be obtained in patients with positive hepatitis B core antibody prior to randomization.
    * Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
  * Active tuberculosis
  * Conditions leading to immune suppression or stimulation of the immune system, such as:

    * Prior treatment with checkpoint inhibitors
    * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided at least 5 half-lives (approximately 75 days) have elapsed since the last dose of anti-CTLA-4 and there was no history of severe immune-mediated adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 or 4)
    * Treatment with systemic immunostimulatory agents (including but not limited to IFN-a, IL-2) for any reason within 6 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment.
    * Prior allogeneic stem cell or solid organ transplant.
* Subjects with a condition requiring systemic treatment with either corticosteroids (≥ 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of randomization/enrollment
* Prior treatment with an anti-DKK1 therapy
* Administration of a live, attenuated vaccine within 30 days prior to the first dose of study medication or anticipation that such a live attenuated vaccine will be required during the study. Any live, attenuated vaccine (e.g. FluMist®) is prohibited while the patient is receiving atezolizumab and for a period of 5 months after discontinuation of atezolizumab. Inactivated influenza vaccines are allowed only during flu season.
* History of osteonecrosis of the hip or evidence of structural bone abnormalities in the proximal femur on magnetic resonance imaging (MRI) scan that is symptomatic and clinically significant. Degenerative changes of the hip joint are not excluded.
* All non hematological toxicities attributed to prior anti-cancer therapy other than hearing loss, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5) or baseline before administration of study drug.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal products.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein; known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Uncontrolled tumor-related pain.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium 1.5 mmol/L, calcium 12 mg/dL or corrected serum calcium ULN)
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina within 3 months prior to initiation of study treatment.

Specific to BTC:

* Ampullary or gallbladder carcinoma
* Patients with liver failure Child-Pugh B or C

Specific to EGC:

• History of hypersensitivity reactions to paclitaxel or other drugs formulated in Cremophor EL (polyoxyethylated castor oil)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months from start of study treatment
  Objective response rate according to RECIST v1.1 is computed as the rate of complete and partial responses (with response confirmation)

SECONDARY OUTCOMES:
Best overall response distribution | 6 months from start of study treatment
  According to RECIST1.1 and iRECIST
Immune objective response rate according to iRECIST | 6 months from start of study treatment
  Immune objective response rate according to iRECIST is computed as the rate of immune complete and partial responses (with response confirmation)
Duration of response using RECIST 1.1 and iRECIST | Until 2 years after start of study treatment
  Response duration will be measured from the time measurement criteria for CR/PR or iCR/iPR are first met until the first date that recurrent or progressive disease is objectively documented, taking as reference the smallest measurements recorded on study (including baseline).
Progression free survival according to RECIST 1.1 and iRECIST | Until 2 years after start of study treatment
  Progression free survival (PFS) according to RECIST 1.1 and iRECIST is defined as the number of days from date of start of treatment to the date of first progression according to RECIST 1.1 or iRECIST respectively or death, whatever comes first. Patients alive and free of progression prior to the analysis cut-off date are censored at the date of the most recent assessment.
Occurrence of adverse events | Until 2 years after start of study treatment
  The study uses the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting
Overall survival (OS) | Until 2 years after start of study treatment
  Overall Survival is defined as the number of days from date of start of treatment to the date of death due to any cause. If a patient has not died, the data will be censored at the last date documented to be alive
Duration of stable disease using RECIST 1.1 and iRECIST | Until 2 years after start of study treatment
  Stable disease duration will be measured from the time of start of treatment until the criteria for progression are met, taking as reference the smallest sum on study (including baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, Study Chair — Universitaetsmedizin - Mainz University Medical Center, Mainz, Germany; Maria Alsina, Study Chair — Vall d'Hebron University Hospital and Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Spain